CLINICAL TRIAL: NCT02457403
Title: A Prospective, Randomized Clinical Trial Comparing Blood Product Use and Bleeding Events During and After Endoscopic or Neurosurgical Procedures in Patients With Cirrhosis and Coagulopathy: Rotational Thromboelastography (ROTEM) Versus Conventional Therapy
Brief Title: Comparison of Blood Product Use and Bleeding Events During and After Endoscopic or Neurosurgical Procedures in Patients With Cirrhosis and Coagulopathy
Acronym: SCARLET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, James Hanje, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2014H0487
Record Dates: First submitted 2015-05-06; First posted 2015-05-29 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-12

CONDITIONS: Cirrhosis; Coagulopathy
MeSH Terms: conditions — Fibrosis; Hemostatic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- ROTEM (Experimental): Transfusion guided by ROTEM during OLT
  Interventions: Device: ROTEM; Other: Conventional Therapy
- Conventional (Active Comparator): Transfusion guided by conventional labs
  Interventions: Device: ROTEM; Other: Conventional Therapy

INTERVENTIONS:
Device: ROTEM — Assess coagulopathy with ROTEM device compared to conventional laboratory tests. ROTEM will be used on all patients, however, determination of blood products used will be based on patient's randomization group.
Other: Conventional Therapy — Assess coagulopathy with conventional laboratory tests (PT/INR, Hemoglobin, Platelet count). Conventional laboratory tests will be obtained on all subjects, however, determination of blood products used will be based on patient's randomization group.

SUMMARY:
A prospective, randomized clinical trial comparing blood product use and bleeding events during and after endoscopic or neurosurgical procedures in patients with cirrhosis and coagulopathy: Rotational Thromboelastometry (ROTEM) vs. conventional therapy (SCARLET).

DETAILED DESCRIPTION:
Orthotopic liver transplantation (OLT) can be associated with significant bleeding requiring multiple blood product transfusions, especially in patients with severe liver dysfunction. Rotational thromboelastometry (ROTEM) is a point-of-care device that has been used successfully to monitor coagulation on whole blood samples during OLT. Whether it allows blood loss and transfusion to be reduced during OLT remains controversial. ROTEM or conventional coagulation tests were used in this study to guide transfusion of platelets, cryoprecipitate, and fresh frozen plasma (FFP) during OLT. Patient characteristics as well as pre- and post- transplant laboratory data were collected. Intra-operative blood loss, type and amount of blood products transfused, and cost were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 and older, admitted to the hospital
* Patients who have clinically documented cirrhosis
* Patients who are coagulopathic (INR > 1.5 and/or platelets < 50,000)
* Patients undergoing an endoscopic procedure or neurosurgical procedure

Exclusion Criteria:

* Patients must not be pregnant
* Patients must not be taking any anticoagulant or antiplatelet medication (with the exception of ASA 81 mg or heparin for DVT prophylaxis)
* Patients must not have an active infection (per PI discretion)
* Patients must not have any known hemostatic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2015-05; Primary Completion 2018-11 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam J Hanje, MD, Principal Investigator — Assistant Professor-Clinical

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a prospective, single center, randomized clinical trial. 34 controls had transfusions guided by conventional labs and 34 participants had transfusions guided by ROTEM during orthotopic liver transplantation.
Groups:
- Conventional: Assess coagulopathy with conventional laboratory tests (PT/INR, Hemoglobin, Platelet count). Conventional laboratory tests will be obtained on all subjects, however, determination of blood products used will be based on patient's randomization group.
Period: Overall Study
Arm/Group | ROTEM | Conventional
Started | 34 (34 participants) | 34 (34 historic controls)
Completed | 34 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ROTEM: Assess coagulopathy with ROTEM device compared to conventional laboratory tests. The ROTEM machine produces values for each of the following: A10-EX, A10-FIB, CT-EX, CT-FIB, and CT-HEP. An algorithm guided the investigator on how to proceed with treatment, whether it be to transfuse 1 unit of platelets & 1 unit of cryo, transfuse 1 unit of cryo, transfuse 1 unit of platelets, transfuse 2 units of platelets, transfuse 2 units fresh frozen plasma (FFP), and whether or not to stop heparin.
- Conventional: Assess coagulopathy with conventional laboratory tests (PT/INR, Hemoglobin, Platelet count, fibrinogen). Based on these lab results, the investigator followed an algorithm and proceeded by either ordering a transfusion of 2 units fresh frozen plasma (FFP), transfusion of 1 unit of platelets, or a transfusion of 2 units of platelets. And if the Fibrinogen came back at < 100 mg/dL, 1 unit of cryoprecipitate was also transfused.
- Total: Total of all reporting groups
Arm/Group | ROTEM | Conventional | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Categorical [Count of Participants; unit: Participants]
  Age: <=18 years | 0 | 0 | 0
  Age: Between 18 and 65 years | 34 | 34 | 68
  Age: >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 21 | 22 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Classified as "white/non-white."
  Participants
    Race/Ethnicity : White | 31 | 31 | 62
    Race/Ethnicity : Non-white | 3 | 3 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34 | 34 | 68
Indication for OLT [Count of Participants; unit: Participants] | 34 | 34 | 68
Model for End-Stage Liver Disease Scale (MELD) score [Mean (Standard Deviation); unit: units on a scale] — MELD score is a scale from 6-40, with a higher score indicating a worse outcome. Population: Raw data was not available so this was the most efficient way to fulfill the "total" column, and there were only 34 participants in each arm.
  units on a scale
    ROTEM: number analyzed (Participants) | 34 | 0 | 34
    ROTEM | 25 (8.37) |  | 25 (8.37)
    Conventional: number analyzed (Participants) | 0 | 34 | 34
    Conventional |  | 22 (7.70) | 22 (7.70)
Presence of hepatocellular carcinoma [Count of Participants; unit: Participants] | 13 | 10 | 23
Presence of portal vein thrombosis [Count of Participants; unit: Participants] | 4 | 2 | 6
Presence of hypercoaguable state [Count of Participants; unit: Participants] | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Intra-operative Blood Loss
Description: Total amount of pre-procedure blood products transfused in patients undergoing endoscopy and neurosurgical procedures.
Time Frame: Patients will be evaluated for the duration of their transfusion (no greater than 24 hour span).
Measure: Median (Inter-Quartile Range); unit: milliliters
Arm/Group | ROTEM | Conventional
Number analyzed (Participants) | 34 | 34
milliliters | 2000 [1500 to 3375] | 3000 [2000 to 7750]

2. Secondary Outcome: Number of Participants With Bleeding Events
Description: Duration of hospitalization is patient dependent, and is not affected by study interventions. Bleeding events (such as post-procedure bleeding, signs/symptoms of bleeding, or active hemorrhage) will be evaluated by chart review for the duration of each subject's hospitalization (up to a maximum of 6 months).
Time Frame: Patients will be assessed for bleeding events from time of consent in the hospital to the time of discharge from the hospitalization (up to a maximum of 6 months).
Measure: Number; unit: participants
Arm/Group | ROTEM | Conventional
Number analyzed (Participants) | 34 | 34
participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Standard definition from clinicaltrials.gov
Arm/Group | ROTEM | Conventional
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT02457403/SAP_000.pdf
  • Study Protocol (2017-01-09): https://cdn.clinicaltrials.gov/large-docs/03/NCT02457403/Prot_001.pdf